CLINICAL TRIAL: NCT02126722
Title: Endofaster Test for Helicobacter Pylori Detection in Patients on Proton Pump Inhibitor Therapy: Prospective Validation
Brief Title: Endofaster Test for Helicobacter Pylori Detection in Patients on Proton Pump Inhibitor Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Niso Biomed S.R.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Helicobacter Infections
Keywords: Helicobacter pylori; Gastritis
MeSH Terms: conditions — Helicobacter Infections; Gastritis | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with dyspepsia on PPI: One hundred patients on PPI will be enrolled among the patients with dyspepsia referred for gastroscopy at Homerton University Hospital. On the day of the endoscopic procedure the patients will bring a stool sample for the detection of faecal Helicobacter pylori antigen. Subsequently, a gastroscopy with multiple biopsies will be performed and during the exam NISO Biomed EndoFaster test, as well as the Clo test, will be carried out.
  Interventions: Procedure: Gastroscopy; Device: EndoFaster test; Other: Clo test; Other: Faecal Helicobacter pylori antigen
- Patients with dyspepsia not on PPI: Fifty patients not on PPI will be enrolled among the patients with dyspepsia referred for gastroscopy at Homerton University Hospital. On the day of the endoscopic procedure the patients will bring a stool sample for the detection of faecal Helicobacter pylori antigen. Subsequently, a gastroscopy with multiple biopsies will be performed and during the exam NISO Biomed EndoFaster test, as well as the Clo test, will be carried out.
  Interventions: Procedure: Gastroscopy; Device: EndoFaster test; Other: Clo test; Other: Faecal Helicobacter pylori antigen

INTERVENTIONS:
Procedure: Gastroscopy — Gastroscopy with multiple biopsies will be performed in all patients enrolled
Device: EndoFaster test — During the gastroscopy the EndoFaster test will be carried out in all patients enrolled.
  Other Names: NISO Biomed EndoFaster test.
Other: Clo test — During the gastroscopy the Clo test will be carried out in all patients enrolled.
Other: Faecal Helicobacter pylori antigen — On the day of the endoscopic procedure all the enrolled patients will bring a stool sample for the detection of Helicobacter pylori antigen.

SUMMARY:
H. pylori infection is the most important causative agent of gastritis, and subsequent atrophic gastritis. The endoscopic diagnosis of H. pylori infection relies on urease tests such as the Clo test. However, treatment with proton pump inhibitors (PPI) impairs the diagnostic yeld of urease tests. The EndoFaster test (NISO BioMed, Turin, Italy) is a new technology that has the advantage, over conventional urease tests, of a real-time analysis of the gastric juice that can provide information regarding Helicobacter pylori infection and pH value of the gastric contents. A well designed clinical study is therefore warranted to fully assess the performance of the EndoFaster test in detecting H. pylori infection in patients treated with PPI. We aim to perform a clinical study in an adult population in United Kingdom in order to determine the diagnostic accuracy of the Endo Faster test compared to the Clo test, histological diagnosis and the faecal antigen test in evaluating H.pylori infection. Patients on PPI will undergo a gastroscopy with multiple biopsies and during the exam NISO Biomed EndoFaster test, as well as the Clo test, will be carried out. H. pylori faecal antigen test will also be performed and used as gold standard. Diagnostic accuracy of the different methods will be determined.

DETAILED DESCRIPTION:
Urease tests such as the Clo test for the diagnosis of Helicobacter pylori infection have been widely used because they are simple, cheap, and easy to carry out (1, 2). They can be performed during the endoscopic exam and give a relatively rapid result. However, treatment with proton pump inhibitors (PPI) may alter the result by changing the milieu where bacteria are present, especially in the antrum, by rendering it inhospitable with consequent decrease in the bacterial load. In addition, PPI themselves may have antiurease properties (3). Another reason for a false-negative result is the presence of intestinal metaplasia (4), which also corresponds to an inhospitable environment for Helicobacter pylori. EndoFaster test is a new technology that has the advantage, over conventional urease tests, of a real-time analysis of the gastric juice that can provide information regarding Helicobacter pylori infection and pH value of the gastric contents. Sensitivity, specificity, PPV and NPV of EndoFaster test for Helicobacter pylori infection resulted to be 98.5%, 87.6%, 84.4% and 98.8 %, respectively. This test may be more accurate than conventional urease tests in the diagnosis of Helicobacter pylori infection in subjects on PPI as indeed it should increase the analysed area, thereby allowing to evaluating the bacterial density in both the gastric antrum and corpus. No data are currently available about the performance of the EndoFaster test in subjects on PPI and a well-designed clinical study is warranted.

The main aim of our study is to conduct a comparative study with the NISO BioMed EndoFaster test, the urease-based test (Clo test), histologic diagnosis and the faecal antigen test (used as the gold standard) for the diagnosis of Helicobacter pylori infection in PPI-treated patients.

We will perform a clinical study using the NISO BioMed Endofaster test to diagnose Helicobacter pylori infection in patients on PPI therapy. The study will be conducted as a collaboration between NISO BioMed (Turin, Italy) and Homerton University Hospital (London, UK). The study will be performed at the Homerton Hospital.

One hundred patients on PPI will be enrolled among the patients with dyspepsia referred for gastroscopy at Homerton University Hospital (London, United Kingdom). A control group of 50 patients with dyspepsia, not on PPI, will be also enrolled in the study.

On the day of the endoscopic procedure the patients will bring a stool sample for the detection of Helicobacter pylori antigen. Subsequently, a gastroscopy with multiple biopsies will be performed and during the exam NISO Biomed EndoFaster test, as well as the Clo test, will be carried out.

Directed biopsies will be collected from the antrum and corpus, following the protocol of the Operative Link for Gastritis Assessment (OLGA) and Sydney classifications for chronic gastritis. Biopsies will be examined at the Pathology laboratory of University College London Hospital and interpreted using the OLGA staging system as well as the Sydney system for the classification of gastritis (5-8).

The performance of the EndoFaster test for the diagnosis of Helicobacter pylori infection will be compared to the Clo test, the histologic diagnosis and the faecal antigen test. In particular, statistical analyses will consist of calculations of the performance indicators of the EndoFaster test, including ROC analysis for cut-off values that give the optimal sensitivity/specificity balance.

The principal goal of this clinical study is to establish the performance of the EndoFaster test in detecting the Helicobacter pylori infection rate in the study population. For this endpoint, we will calculate sensitivity (SE), specificity (SP), negative predictive value (NPV), positive predictive value (PPV) and AUC (area under ROC curve), collectively and individually for each 4 tests. ROC analysis can be used to estimate the best SE/SP balance for each single test. One of the aims is to establish the best cut-offs in order to give the EndoFaster test an optimal performance.

Additionally, clinically significant conditions (gastric atrophy, intestinal metaplasia, gastric cancer) will be recorded and the association rate with Helicobacter pylori infection will be studied (9,10).

The necessary preparations for the study execution at Homerton University Hospital NHS Foundation Trust will start immediately when the hospital has reached the agreement with NISO BIOMED. The study plan necessitates a review by the institutional review board (IRB, Ethical Committee) before permission to start.

We aim to obtain unbiased (i.e., 100% confirmed by the gold standard, i.e. faecal antigen test) estimate for the performance of EndoFaster test in detecting the Helicobacter pylori infection rate in patients on PPI treatment. This will include determining the optimal cut-offs that give the optimal SE/SP balance for detecting the study endpoint. Application of these cut-offs in clinical practice would lead to optimised performance of EndoFaster test.

ELIGIBILITY:
Inclusion Criteria:

* Adult females and males over 45 years of age with dyspeptic symptoms (epigastric pain, bloating and epigastric discomfort)

Exclusion Criteria:

* Patients who require surgery or immediate follow-up treatment for major symptoms, including hematemesis, melena, acute epigastric pain
* Patients who previously underwent upper gastrointestinal surgery
* Patients with diabetes
* Pregnant women
* Subjects who refuse to participate or are unable to give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients on PPI will be enrolled among the patients with dyspepsia referred for gastroscopy at Homerton University Hospital (London, United Kingdom). A control group of 50 patients with dyspepsia, not on PPI, will be also enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the EndoFaster test in H. pylori diagnosis | Six weeks
  Clinical specialist consultation will be performed and eligible patients will be enrolled and candidate to undergo a gastroscopy.
  On the day of the endoscopic procedure the patients will bring a stool sample for the detection of Helicobacter pylori antigen. Subsequently, a gastroscopy with multiple biopsies will be performed and during the exam NISO Biomed EndoFaster test, as well as the Clo test, will be carried out.
  Performance indicators (sensitivity, specificity, positive predictive value, PPV, negative predictive value, NPV and their 95%CI) of the EndoFaster test will be calculated, using the STATA/SE software. The area under ROC (Receiver Operating Characteristics) called AUC, will be identified. These ROC curves can be used to identify the optimal sensitivity/specificity balance that gives each biomarker an optimal threshold for detection of each study endpoint. Significance of the difference between AUC values can be estimated using STATA's roccomb test with 95%CI.

CONTACTS AND LOCATIONS:
Overall Officials: Cinzia Papadia, MD, Principal Investigator — Homerton University Hospital; Ray Shidrawi, MD, Study Director — Homerton University Hospital; Marco Novelli, MD, Study Chair — University College, London
Locations (1):
- Homerton University Hospital, London, United Kingdom